CLINICAL TRIAL: NCT07355634
Title: A Randomized, Placebo-Controlled Trial Evaluating the Impact of a Synbiotic Dietary Supplement on Markers of Gastrointestinal Health
Brief Title: Terraflora Daily Care and Gastrointestinal Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OvationLab (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ENV-001
Record Dates: First submitted 2026-01-02; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Terraflora - Daily Care (Experimental)
  Interventions: Dietary Supplement: Synbiotic Dietary Supplement
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic Dietary Supplement — 12 weeks of supplementation with Enviromedica - Terraflora Daily Care
  Arms: Terraflora - Daily Care
Dietary Supplement: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
A 12-week, randomized, double-blind, placebo-controlled clinical trial will be conducted evaluating the effectiveness of Enviromedica - Terraflora Daily Care on markers of gastrointestinal function and symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females age ≥ 25 years
2. Ability to read and speak English
3. Dysbiosis (≥3 on GA-Map Dysbiosis Score) on a stool test (GI360 Profile, Doctor's Data, St. Charles, Illinois)

Exclusion Criteria:

1. Daily use within the past month of any probiotic or prebiotic supplement
2. Current diagnosis of inflammatory bowel disease, including Crohn's or ulcerative colitis
3. Current daily usage of non-steroidal anti-inflammatory drugs (NSAID), proton pump inhibitors (PPI), or antibiotic medications
4. Current daily tobacco smoker
5. Known allergies to any substance in the study products
6. Currently pregnant or lactating women or women planning to become pregnant in the next 12 weeks
7. Current diagnosis of any other chronic health condition (e.g., cancer, chronic kidney disease) deemed clinically contraindicated for the study protocol
8. Current participation in another clinical trial
9. Participants unable to provide consent

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
GA-Map Dysbiosis Test | 4 weeks, 12 weeks

SECONDARY OUTCOMES:
Percentage of participants with dysfunction on GI360 Profile | 4 weeks, 12 weeks
Percentage of participants with dysfunction on Thorne Gut Health Test | 4 weeks, 12 weeks
Gastrointestinal Symptom Rating Scale | 4 weeks, 12 weeks
  Minimum value: 1, Maximum value: 7, Higher scores represent more severe/troublesome symptoms.

IPD SHARING:
Plan to Share IPD: No